CLINICAL TRIAL: NCT00152087
Title: Treatment of Unresectable Hepatocellular Carcinoma With Therasphere. A Human Device Evaluation Protocol.
Brief Title: A Non-Randomized Study of Internal Radiation Therapy to the Liver in Patients With Primary Liver Cancer for Whom Surgery is Not Possible.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Hospital, Florida (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJCI015; Alison Calkins, MD; Matthew Berlet, MD
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2005-09-09 (Estimated); Status verified 2005-09

CONDITIONS: Liver Cancer
Keywords: Liver cancer; Brachytherapy
MeSH Terms: conditions — Liver Neoplasms | interventions — Brachytherapy

INTERVENTIONS:
Device: Brachytherapy

SUMMARY:
Surgical resection of the affected liver offers the best chance for disease-free survival in patients with Hepatoma (HCC). Unfortunately, most hepatoma patients present with disease which is multi-focal and thus not resectable. Fewer than 15% of HCC patients are resectable. The objective of treatment with TheraSphere is to selectively administer a dose of radioactive material directly to neoplastic tissue in the liver. Systemic therapy is largely ineffective.

DETAILED DESCRIPTION:
Protocol Objectives include:

* Determine the proportion of patients with HCC in whom the treatment plan can be completed
* Evaluate the response to therapy
* Evaluate toxicities and adverse experiences associated with TheraSphere treatment
* Evaluate survival time

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age of any sex, race
* Histological proof of HCC
* Able to give Informed Consent
* ECOG performance equal or less than 2
* Life expectancy equal to or greater than 3 months
* Non- pregnant with acceptable contraception in premenopausal women
* Greater than 4 weeks since prior radiation therapy or surgery
* 1 month post chemotherapy
* Serum Bilirubin < 2.0
* Acceptable white blood count

Exclusion Criteria:

* Co-morbid disease that would place patient at undue risk.
* Pre-existing diarrhea/illness
* Pregnant
* Fail preliminary MAA testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2002-10; Study Completion 2005-06

PRIMARY OUTCOMES:
Efficacy
- Response to treatment
- Survival time from treatment
Safety:
- Adverse experience

CONTACTS AND LOCATIONS:
Overall Officials: Alison R. Calkins, MD, Principal Investigator — St. Joseph's Hospital, Tampa, FL
Locations (1):
- St. Joseph's Hospital, Tampa, Florida, United States

REFERENCES:
- See also: St Joseph's Hospital web site — http://www.sjbhealth.org